CLINICAL TRIAL: NCT03947632
Title: Anthropometric Measurements in Children Having Transfusion-dependent Beta Thalassemia.
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Bushra Moiz, Professor, Aga Khan University
Other Study IDs: 2305-Pat-ERC-12
Record Dates: First submitted 2019-05-07; First posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Beta Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Five milliliter of blood samples were collected in two tubes (ethylenediaminetetraacetic acid and gel)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum ferritin and hemoglobin test — Five milliliter of blood samples were collected in two tubes (ethylenediaminetetraacetic acid and gel) at Fatimid foundation by a trained phlebotomist prior to blood transfusion to determine hemoglobin and serum ferritin.

SUMMARY:
The aim of this study was to determine the anthropometric measurements in transfusion-dependent β-thalassemia children in Pakistan. The secondary aim was to correlate serum ferritin with the physical growth

DETAILED DESCRIPTION:
Material and methods

Setting The study was conducted at the Sections of Hematology and Clinical Chemistry in the Department of Pathology and Laboratory Medicine, Aga Khan University, Karachi, Pakistan during January 2013 to December 2014. Patient recruitment was conducted at a non-profit organization named Fatimid Foundation Karachi (FFK), which provides free of cost blood components to the patients with various blood disorders. There are more than 4000 registered patients of thalassemia and hemophilia at FFK.

Patient selection After informed consent from their parents, 367 pediatric patients (age 5-17 year) with transfusion-dependent β-thalassemia were recruited. All patients were diagnosed based on hemoglobin electrophoresis or high-performance liquid chromatography.

Data collection Detail history was collected by a trained research officer on a predetermined questionnaire. The following information was collected from medical records of the patients: demographics (age, gender, age at the time of diagnosis and at first transfusion), anthropometrics (height and weight), and clinical details (blood transfusion history, iron chelation, last pre-transfusion hemoglobin, and last serum ferritin levels).

Sample collection Five milliliter of blood samples were collected in two tubes (ethylenediaminetetraacetic acid and gel) at Fatimid foundation by a trained phlebotomist prior to blood transfusion to determine hemoglobin and serum ferritin.

Laboratory methodology Serum ferritin was measured by chemi-luminescent micro-particle immunoassay on Cobos® E-601 and hemoglobin was measured using Sysmex® XP-100.

Anthropometry World health organization (WHO) 2007 growth charts were used for boys and girls to assess their physical growth. Body mass index (BMI) was computed as weight in kg/height in square meters. z-Score of height (h-SDS), weight (w-SDS) and BMI. According to WHO reference 2007, a z-score of <-2 for height was considered as stunted growth and BMI of <-2 was considered as underweight or thin for age.

Statistical analysis Data were collected, managed, edited, entered, and analyzed by statistical package of social sciences (SPSS) version 22 and STATA 13 (Stata Corp, College Station, TX, U.S.A.). A descriptive analysis of all patients in the study was performed. In order to analyze the profile of the sample according to the variables studied, frequency tables for categorical variables like (gender, age group) were created. Male: female ratio was also computed. The mean ± standard deviation, minimum and maximum values were calculated for parametric and median and interquartile range (IQR; Q3-Q1) for non-parametric variables. Spearman rho correlation was used to test relationships between the non-parametric variables. The level of significance taken for all the statistical tests was a p-value of <0.05. The association of h-SDS with median serum ferritin levels was further confirmed by comparing these laboratory parameters in children with height z-scores <2 with those with the z-score ≥2 using the Mann-Whitney test.

ELIGIBILITY:
Inclusion Criteria:

* Children with transfusion dependent beta thalassemia major
* Age 5 to 17 years
* Subjects with informed consent

Exclusion Criteria:

* Age more than 17 years
* Subjects who refused informed consent

Ages: 5 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: 367 pediatric patients (age 5-17 year) with transfusion dependent β-thalassemia were recruited. All patients were diagnosed based on hemoglobin electrophoresis or high-performance liquid chromatography. Patient recruitment was conducted at a non- profit organization named Fatimid Foundation Karachi (FFK), which provides free of cost blood components to the patients with various blood disorders.
Sampling Method: Non-Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Height in transfusion-dependent β-thalassemia pediatric patients in Pakistan were recorded to assess growth rate | Jan 2013 to Dec 2014
  Height in meters will be recorded from medical records of the patients
Weight in transfusion-dependent β-thalassemia pediatric patients in Pakistan were recorded to assess growth rate | Jan 2013 to Dec 2014
  Wight in kilograms will be recorded from medical records of the patients
Assessment of physical growth in transfusion-dependent β-thalassemia pediatric patients in Pakistan were recorded to assess growth rate | Jan 2013 to Dec 2014
  World health organization (WHO) 2007 growth charts were used for boys and girls to assess their physical growth. Body mass index (BMI) was computed as weight in kg/height in square meters (kg/m^2). z-Score of height (h-SDS), weight (w-SDS), and BMI (BMI-SDS) were also calculated.
Serum ferritin levels and their association with z-Score of height | Jan 2013 to Dec 2014
  Correlation was assessed between height for age z-score and serum ferritin levels. Serum ferritin was measured by chemi-luminescent micro-particle immunoassay on Cobos® E-601. The association of z-Score of height with median serum ferritin levels was further confirmed by comparing these laboratory parameters in children with height z-scores <2 with those with the z-score ≥2 using the Mann-Whitney test.

IPD SHARING:
Plan to Share IPD: No